CLINICAL TRIAL: NCT07274215
Title: Impact of Intraoperative Paragastric Block on Visceral Pain and Postoperative Nausea and Vomiting After Sleeve Gastrectomy: A Randomized Controlled Trial
Brief Title: Paragastric Block for Pain and PONV in Sleeve Gastrectomy
Acronym: BLOCK-SG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Abdullah Sisik, Professor of General Surgery, Istanbul Gedik University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 186123-20.06.2025
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Nausea and Vomiting; Postoperative Pain After Laparoscopic Sleeve Gastrectomy
Keywords: postoperative pain; postoperative nausea and vomiting; VAS; sleeve gastrectomy; paragastric block
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned in a 1:1 ratio to one of two parallel groups: (1) intraoperative paragastric block with 0.5% bupivacaine or (2) sham block with isotonic saline. Each participant will receive only one type of intervention throughout the study. No crossover will occur between groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgical team, anesthesia providers, patients, data collectors, and outcome assessors will all remain blinded to group allocation. To preserve masking, both the intervention and placebo procedures will be performed identically in terms of injection site, volume, and technique. Group assignment will be concealed using sequentially numbered, opaque envelopes opened only after induction of anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paragastric Block with Bupivacaine (Experimental): Participants in this group will undergo laparoscopic sleeve gastrectomy with intraoperative paragastric block. A total of 20 mL of 0.5% bupivacaine will be injected into six predefined anatomical sites around the stomach under direct laparoscopic visualization after gastric resection. The block targets autonomic nerve plexuses to reduce postoperative visceral pain and nausea. The injection will be performed using a standardized technique with a 25G needle.
  Interventions: Drug: Bupivacaine 0.5%
- Sham Block with Isotonic Saline (Placebo Comparator): Participants in this group will undergo laparoscopic sleeve gastrectomy with a sham paragastric block. A total of 20 mL of isotonic saline will be injected into the same six anatomical sites using the same technique, timing, needle type, and volume as the intervention group, ensuring proper blinding. No active local anesthetic will be used.
  Interventions: Drug: Isotonic Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Bupivacaine 0.5% — Participants receive 20 mL of 0.5% bupivacaine administered intraoperatively as a paragastric block. The injection is performed under laparoscopic guidance at six predefined anatomical sites around the stomach following gastric resection.
  Arms: Paragastric Block with Bupivacaine
Drug: Isotonic Saline (0.9% NaCl) — Participants receive 20 mL of isotonic saline (placebo) administered intraoperatively using the same injection technique and anatomical landmarks as the active treatment group, to maintain blinding.
  Arms: Sham Block with Isotonic Saline

SUMMARY:
This single-center, prospective, randomized, double-blind controlled trial aims to evaluate the effects of intraoperative paragastric block (PGBLOCK) on early postoperative visceral pain, postoperative nausea and vomiting (PONV), and analgesic requirements in patients undergoing laparoscopic sleeve gastrectomy (LSG). Despite advancements in multimodal analgesia protocols, visceral pain remains a significant postoperative concern following LSG, contributing to increased opioid use and delayed recovery. Paragastric block is a novel technique targeting autonomic neural pathways-such as branches of the celiac ganglia and vagal nerves-through precise intraoperative injection of local anesthetics near the stomach.

A total of 180 patients scheduled for elective LSG will be randomized in a 1:1 ratio to receive either paragastric block with 20 mL of 0.5% bupivacaine or a sham block with 20 mL of isotonic saline. Injections will be administered at six predefined anatomical sites under laparoscopic guidance after gastric resection. The surgical technique, anesthetic protocol, and postoperative care will be standardized for all participants. Both patients and clinical personnel involved in care and outcome assessment will remain blinded to group assignment.

The primary outcome is the assessment of postoperative visceral pain using Visual Analog Scale (VAS) scores at 0 and 2 hours postoperatively. Secondary outcomes include PONV severity grading, mobilization status, total analgesic consumption (pethidine + tramadol), and need for rescue antiemetics within the first 24 hours post-surgery. Exclusion criteria include history of upper abdominal surgery, chronic opioid use, pregnancy, severe systemic disease, or allergy to medications used in the protocol.

This study is expected to provide high-quality evidence regarding the efficacy of paragastric block in improving early postoperative recovery and reducing opioid reliance after LSG.

DETAILED DESCRIPTION:
Introduction Laparoscopic sleeve gastrectomy (LSG) is one of the most frequently preferred methods for surgical treatment of obesity. However, postoperative visceral pain and its associated autonomic manifestations, particularly postoperative nausea and vomiting (PONV), significantly impair patient recovery, delay mobilization, and extend hospitalization duration. Contemporary multimodal analgesia protocols effectively address somatic components of pain but demonstrate limited efficacy in managing visceral pain pathways, which predominate following LSG. This results in increased opioid use and related complications. Paragastric block (PGBLOCK) represents an emerging technique specifically designed to target the autonomic neural pathways responsible for visceral pain transmission. This technique involves precise infiltration of local anesthetics to autonomic nerve plexuses surrounding the stomach, including branches of the celiac ganglia and vagal pathways.

This study was designed to evaluate the effects of intraoperative paragastric block application on early postoperative visceral pain, PONV, and analgesic requirements in patients undergoing LSG.

Materials and Methods Study Design This study will be designed as a single-center, prospective, randomized, controlled, double-blinded clinical trial. This study will comply with both the ethical standards of the institutional and/or national research committee and the principles outlined in the 1964 Helsinki Declaration and its later amendments. The study protocol will be reviewed and approved by the Ethics Committee of Marmara University School of Medicine. Following the approval of the ethics committee, the study will be registered at ClinicalTrials.gov.

A total of 180 patients will be randomized into two groups: the intervention group undergoing LSG with intraoperative paragastric block using 20 mL of 0.5% bupivacaine (n=90), and the placebo group undergoing LSG with sham paragastric block using 20 mL of isotonic saline (n=90). In both groups, the injection will be performed at six predefined anatomical sites under direct laparoscopic visualization, following completion of gastric resection. To preserve blinding, the procedural technique-including injection sites, needle type, and volume-will be identical in both groups. Neither the surgical team nor the patients will be aware of the group allocation. The study will include a CONSORT flow diagram illustrating participant progression through all trial phases.

Inclusion Criteria

* Patients aged between 18 and 65 years.
* Candidates scheduled for elective LSG.
* American Society of Anesthesiologists (ASA) physical status classification I-III.
* Ability to provide written informed consent and willingness to comply with study procedures.

Exclusion Criteria

* History of prior upper abdominal surgery.
* Known psychiatric or neurological disorders that could interfere with pain assessment or postoperative care.
* History of opioid dependency or chronic opioid use.
* Allergy or hypersensitivity to local anesthetics or any of the medications used in the study protocol (e.g., paracetamol, dexketoprofen, ondansetron, tramadol, metoclopramide).
* Severe hepatic, renal, or cardiac dysfunction (e.g., cirrhosis, end-stage renal disease, heart failure).
* Pregnancy or breastfeeding.
* Concomitant surgery (e.g., cholecystectomy, hiatal hernia repair, or abdominal wall repair).
* Known bleeding disorders or coagulopathy (e.g., INR >1.5, platelet count <50,000/mm³, or ongoing anticoagulant therapy)

Randomization and Blinding After obtaining informed consent, eligible patients will be randomized in a 1:1 ratio into either the block group or the control group using a computer-generated randomization sequence. Allocation will be implemented using sequentially numbered, sealed opaque envelopes prepared by an independent researcher not involved in the study. To ensure allocation concealment, the envelope will be opened only after the induction of anesthesia.

This study is double-blinded: both the patients and all clinical personnel involved in intraoperative care, postoperative follow-up, data collection, and outcome assessments will remain unaware of group assignments throughout the study to minimize performance and detection bias.

Anesthesia Protocol General anesthesia will be induced intravenously without premedication after establishing standard monitoring. Anesthesia will be induced with intravenous propofol (2.5-3.5 mg/kg), fentanyl (1 μg/kg), and rocuronium bromide (0.6 mg/kg). Maintenance of anesthesia will be provided with 2% sevoflurane and 100% oxygen, with remifentanil infusion at a dose of 0.1-0.4 μg/kg/min during the intraoperative period.

All patients will receive intravenous paracetamol (1,000 mg) and dexketoprofen trometamol (50 mg) intraoperatively. These agents will be continued intravenously in the postoperative period as part of the routine analgesia protocol at 6-hour and 8-hour intervals, respectively.

Upon arrival to the recovery unit (designated as hour 0), all patients will receive intravenous pethidine (100 mg). In cases where the Visual Analog Scale (VAS) score is ≥4, intravenous tramadol (100 mg) will be administered as rescue analgesia when necessary.

For PONV prophylaxis, intravenous ondansetron (8 mg) will be administered intraoperatively. Patients who develop nausea and/or vomiting in the postoperative period will receive intravenous metoclopramide (10 mg) as rescue antiemetic.

Surgical Technique All laparoscopic sleeve gastrectomy (LSG) procedures will be performed under general anesthesia by two experienced bariatric surgeons (Dr. H.E. and Dr. A.Ş.) using a standardized five-port technique. After establishing pneumoperitoneum at 12-14 mmHg by direct insertion of the camera trocar, the greater curvature of the stomach will be mobilized, starting 4-6 cm proximal to the pylorus and continuing up to the angle of His. Dissection of the gastrocolic, gastrosplenic, and posterior attachments will be performed using a LigaSure™ vessel sealing device (Medtronic, USA). Gastric resection will be performed using sequential applications of a linear stapler, calibrated by a 36 French bougie positioned along the lesser curvature. Oversewing of the staple line with 3-0 PDS sutures and omentopexy will be performed in all patients. In both groups, the study injection (block or placebo) will be administered prior to oversewing and omentopexy, in accordance with the group assignment.

Paragastric Block Procedure After completion of gastric resection, paragastric autonomic nerve blockade will be performed by injecting a total of 20 mL of 0.5% bupivacaine into six separate points: along the lesser curvature around the left gastric artery using a 25G needle guided by laparoscopic visualization. In the control group, an identical procedure will be performed using 20 mL of isotonic saline (SF) to maintain blinding. Both the surgical team and the patients will remain blinded to the solution administered.

Postoperative Care and Follow-up All patients will be transferred to the postoperative care unit after completion of surgery.

Routine postoperative analgesia will include intravenous paracetamol (1 g every 6 hours) and dexketoprofen trometamol (50 mg every 8 hours). Rescue analgesia with intravenous tramadol (100 mg) will be administered if the VAS score is ≥4.

For antiemetic prophylaxis, intravenous ondansetron (8 mg) will be routinely administered intraoperatively. In cases of postoperative nausea and/or vomiting, intravenous metoclopramide (10 mg) will be administered as a rescue antiemetic.

Postoperative evaluations will be performed at 0, 2, 6, and 12 hours post-surgery, including assessment of VAS scores, PONV grading scale, and mobilization status. VAS scores will be measured on a 10-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). PONV severity will be evaluated using a standardized grading scale as follows:

* Grade 0: No nausea or vomiting.
* Grade 1: Nausea without vomiting.
* Grade 2: Nausea accompanied by vomiting fewer than three times per day (<3 times/day).
* Grade 3: Vomiting three or more times per day (≥3 times/day). All patients will be followed up until 24 hours postoperatively for outcome assessment and analgesic/antiemetic requirement recording.

Endpoints

The following variables will be evaluated in the study:

* Primary endpoint:

  o VAS scores at hours 0 and 2
* Secondary endpoints:

  * PONV grades at hours 0 and 2
  * VAS and PONV grades at hours 6 and 12
  * Early mobilization status at hour 2
  * Total analgesic requirement in the first 24 hours (pethidine + tramadol consumption)
  * Rescue antiemetic requirement

Statistical Analysis Statistical analyses will be performed using SPSS for Windows version 26.0 (IBM Corp., Armonk, NY, USA). The normality of the distribution of continuous variables will be evaluated using the Kolmogorov-Smirnov and Shapiro-Wilk tests. Continuous variables will be expressed as mean ± standard deviation (SD) for normally distributed data and as median (interquartile range [IQR]) for non-normally distributed data.

For the comparison of continuous variables between the two groups, the independent samples t-test will be used for normally distributed data, and the Mann-Whitney U test will be used for non-normally distributed data. Categorical variables will be presented as numbers and percentages, and comparisons between groups will be performed using the chi-square test or Fisher's exact test where appropriate. A two-tailed p-value <0.05 will be considered statistically significant.

Sample Size Calculation A power analysis was performed to determine the number of patients required for the study. Based on the data reported in the article titled "Paragastric Autonomic Neural Blockade to Prevent Early Visceral Pain and Associated Symptoms After Laparoscopic Sleeve Gastrectomy: a Randomized Clinical Trial" by Daes et al., the effect size (Cohen's d) was calculated as 0.744. To achieve a 95% confidence level (α = 0.05) and 95% power (β = 0.05), the minimum required sample size was determined to be 106 patients (53 per group). Considering potential dropouts, a total of 180 patients were included. Power analysis was performed using G*Power version 3.1 , Heinrich-Heine-University Düsseldorf, Germany.

ELIGIBILITY:
Inclusion Criteria

* Patients aged between 18 and 65 years.
* Candidates scheduled for elective LSG.
* American Society of Anesthesiologists (ASA) physical status classification I-III.
* Ability to provide written informed consent and willingness to comply with study procedures.

Exclusion Criteria

* History of prior upper abdominal surgery.
* Known psychiatric or neurological disorders that could interfere with pain assessment or postoperative care.
* History of opioid dependency or chronic opioid use.
* Allergy or hypersensitivity to local anesthetics or any of the medications used in the study protocol (e.g., paracetamol, dexketoprofen, ondansetron, tramadol, metoclopramide).
* Severe hepatic, renal, or cardiac dysfunction (e.g., cirrhosis, end-stage renal disease, heart failure).
* Pregnancy or breastfeeding.
* Concomitant surgery (e.g., cholecystectomy, hiatal hernia repair, or abdominal wall repair).
* Known bleeding disorders or coagulopathy (e.g., INR >1.5, platelet count <50,000/mm³, or ongoing anticoagulant therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Visceral pain score measured by Visual Analog Scale (VAS) | At 0 and 2 hours postoperatively
  Postoperative visceral pain will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Scores will be recorded by blinded observers at specific postoperative time points.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) grade | At 0, 2, 6, and 12 hours postoperatively
  PONV will be evaluated using a standardized 4-point grading scale: Grade 0 (no nausea/vomiting), Grade 1 (nausea only), Grade 2 (nausea with <3 vomiting episodes/day), Grade 3 (≥3 vomiting episodes/day).
Cumulative analgesic consumption (pethidine + tramadol) | Within 24 hours postoperatively
  Total dose of rescue analgesics (pethidine and tramadol) administered during the first 24 hours after surgery will be recorded in milligrams for each patient.
Rescue antiemetic requirement | Within 24 hours postoperatively
  Use of rescue antiemetic medication (metoclopramide 10 mg IV) will be recorded if postoperative nausea or vomiting occurs despite prophylactic ondansetron.
Early mobilization status | At 2 hours postoperatively
  Patient mobilization (defined as sitting upright or ambulating) will be assessed at 2 hours postoperatively and documented as "mobilized" or "not mobilized."

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gedik University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01 October 2025- 01 December 2025